CLINICAL TRIAL: NCT01139424
Title: Safety and Efficacy of Closure of Postoperative Anastomotic Leaks in the Stomach and Esophagus by Endoscopic Suturing: A Prospective Pilot Study
Brief Title: Closure of Anastomotic Leaks in the Stomach and Esophagus by Endoscopic Suturing
Acronym: GASTROSUTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Professor Fritscher-Ravens, UKSH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-Fritscher-Ravens; UKSH1 (Other: UKSH)
Record Dates: First submitted 2010-05-28; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-05

CONDITIONS: Postoperative; Anastomosis, Surgical
Keywords: surgical leak; endoscopic suturing; Anastomotic leakage; esophageal or gastric resection
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label treatment arm (Experimental): endoscopic suturing
  Interventions: Device: endoscopic suturing

INTERVENTIONS:
Device: endoscopic suturing — endoscopic suturing of the anastomotic leak
  Other Names: Using the Ethicon Endosurgery InScope tissue apposition system (TAS).; FDA regulation number 21 CFR 876.1500, CE#: CE0123 (G2S 09 12 57666 029)

SUMMARY:
Patients with suspected leakage at the specified surgical anastomoses undergo an immediate diagnostic endoscopy as part of current clinical routine. Consenting patients meeting the inclusion criteria will undergo closure of the defect by endoscopic suturing in addition to standard surgical care.

ELIGIBILITY:
Inclusion Criteria:

* leakage at anastomosis within 2 weeks after upper gastrointestinal (GI) resection

Exclusion Criteria:

* tubular ischemia of the upper GI tract
* inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety | 2 years
  Endpoint to be recorded during hospital stay: Composite serious adverse event endpoint for 30 days after the diagnosis of anastomotic leakage including:
  * Death
  * Injury to vessels through the suture device, leading to bleeding or thrombosis
  * Cardiac tamponade, arrhythmia
  * Pneumothorax
  * Bleeding requiring transfusion
  * possible medium-term complications such as new mediastinal abscess
Technical feasibility | 2 years
  Technical success of the anastomotic closure

SECONDARY OUTCOMES:
Time to healing of the anastomotic leak | 2 years
  Scored during the hospital stay until 6 months after the original operation. Patients who die or undergo complete resection of the organ (e. g. esophagectomy with cervical fistula) are scored as "nevel healed" - i.e. censored events. Efficacy statistics need to use local historic controls and literature data. Statistical analysis will be performed using the LogRank test.
Long term safety | 6 months after diagnosis of anastomotic leakage
  Long term safety
  * Anastomotic stenosis, as assessed by endoscopy
  * Clinically apparent functional problems (e.g. dysphagia, incontinence)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Fritscher-Ravens, MD, Principal Investigator — UKSH
Locations (1):
- UKSH, Kiel, Schleswig-Holstein, Germany